CLINICAL TRIAL: NCT07377123
Title: Application of Tubeless Spontaneous Ventilation Anesthesia in Kidney Transplantation Surgery: A Single-Center, Prospective, Randomized Controlled Trails
Brief Title: Tubeless Spontaneous Ventilation Anesthesia in Kidney Transplantation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jianxing He (Other)
Responsible Party: Sponsor-Investigator, Jianxing He, Clinical Professor, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ES-2025-130-02
Record Dates: First submitted 2025-12-04; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Kidney Transplantation; CKD (Chronic Kidney Disease) Stage 5D
Keywords: kidney transplantation; tubeless; ERAS; anesthesia
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: This study is designed as a single-center, prospective, randomized controlled clinical trial. Patients awaiting kidney transplantation at our hospital will be the study subjects and included in the study according to the inclusion/exclusion criteria. Using a block randomization method, two kidney transplant patients receiving kidneys from the same donor will be randomly assigned to the experimental group and the control group.
  Experimental Group: Tubeless spontaneous ventilation anesthesia (TSVA) Control Group: Endotracheal tube anesthesia (ETT) The two groups will be compared in terms of anesthetic drug dosage (dosage of muscle relaxants, anesthetic analgesics, and sedatives), anesthetic effect and intraoperative ventilation effect, intraoperative hemodynamics, surgery/anesthesia duration; postoperative awakening recovery time; perioperative patient pain scores; postoperative pulmonary complications and non-pulmonary complications, recovery of transplanted kidney function etc.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tubeless Spontaneous Ventilation Anesthesia (TSVA) (Experimental)
  Interventions: Procedure: Tubeless Spontaneous Ventilation Anesthesia
- Endotracheal Tube Anesthesia (ETT) (Active Comparator)
  Interventions: Procedure: Endotracheal Tube Anesthesia

INTERVENTIONS:
Procedure: Tubeless Spontaneous Ventilation Anesthesia — 1. Pre-anesthesia induction: Midazolam 2-3 mg intravenous injection.
  2. Laryngeal mask insertion: After spontaneous breathing stabilizes, select an appropriate size laryngeal mask for insertion.
  3. Anesthesia depth monitoring: Maintain Bispectral Index (BIS): 40-60.
  4. Anesthesia induction and maintenance: Continuous intravenous infusion of Propofol 0.5-2.0 mg/ml (TCL mode), Dexmedetomidine.
  5. Analgesia: Sufentanil initial dose, Remifentanil maintenance analgesia.
  6. Muscle relaxant: Cisatracurium initial dose 2-10 mg, to reduce abdominal muscle tension without excessively suppressing spontaneous breathing. Additional doses may be given during surgery based on the situation.
  7. Intraoperative monitoring: Continuous monitoring of ECG, heart rate, invasive blood pressure, SpO₂; intermittent monitoring of end-tidal CO₂, tidal volume, fraction of inspired oxygen during airway patency; regular arterial blood gas analysis.
  Arms: Tubeless Spontaneous Ventilation Anesthesia (TSVA)
Procedure: Endotracheal Tube Anesthesia — 1. Pre-anesthesia induction, anesthesia maintenance, and analgesic medication are consistent with the TSVA group.
  2. Muscle relaxant: Conventional protocol (induction dose: 0.2 mg/kg, supplemental dose: 4-6 mg every 40 minutes). Additional muscle relaxants are intermittently administered later based on intraoperative muscle relaxation effect and patient response to stimulation.
  3. After successful endotracheal intubation, connect to the anesthesia machine for continuous mechanical ventilation (tidal volume 6-8 ml/kg).
  4. Anesthesia depth monitoring: Maintain Bispectral Index (BIS): 40-60.
  5. Intraoperative monitoring: Continuous monitoring of ECG, heart rate, invasive blood pressure, SpO₂; intermittent monitoring of end-tidal CO₂, tidal volume, fraction of inspired oxygen during airway patency; regular arterial blood gas analysis.
  Arms: Endotracheal Tube Anesthesia (ETT)

SUMMARY:
The aim of this clinical trial is to compare the intraoperative use of neuromuscular blocking agents and other anesthetic drugs between tubeless spontaneous ventilation anesthesia (TSVA) and conventional endotracheal intubation (ETT) anesthesia in kidney transplantation. The study will also evaluate the safety, stability, and postoperative recovery associated with TSVA.

This trial is designed to address the following questions:

* Does TSVA reduce the intraoperative requirement for neuromuscular blocking agents and other anesthetic medications?
* Does TSVA improve postoperative outcomes in kidney transplant recipients?
* How do the intraoperative safety and stability of TSVA compare with those of ETT anesthesia?

Researchers will compare anesthetic drug consumption, intraoperative anesthetic performance, and postoperative recovery outcomes between the TSVA and ETT groups to determine whether TSVA can decrease anesthetic drug use and enhance patient recovery.

Participants will:

* Undergo a complete preoperative assessment
* Receive kidney transplantation under TSVA or ETT anesthesia, with relevant intraoperative data recorded
* Receive tubeless postoperative management, with documentation of pain scores, complications, and recovery of graft function
* Be followed throughout their lifetime after discharge, providing long-term follow-up information

ELIGIBILITY:
Inclusion Criteria:

1. No gender restriction, age 18-65 years (including upper and lower limits).
2. First-time recipient of citizen organ donation kidney transplantation.
3. Type of citizen organ donation must be Category I China (Donation after Brain Death DBD).
4. Donor and recipient blood type identical.
5. Panel reactive antibody (PRA) results negative within six months preoperatively.
6. Body mass index (BMI) <28 kg/m².
7. No severe pulmonary ventilation or gas exchange dysfunction, preoperative pulmonary function assessment meets kidney transplantation requirements, preoperative chest CT shows no significant abnormalities.
8. No severe arrhythmia (frequent atrial fibrillation or ventricular premature beats), normal cardiac function (ejection fraction > 50%).
9. American Society of Anesthesiologists (ASA) physical status classification ≤ III.
10. Voluntarily participate in clinical research, fully understand this study and voluntarily sign the informed consent form, and complete all trial procedures.

Exclusion Criteria:

1. Combined multi-organ transplantation.
2. Previous history of organ transplantation other than kidney.
3. Living donor kidney transplantation.
4. If one of the two patients receiving a kidney from the same donor does not meet the inclusion criteria, the other patient is also excluded.
5. Previous history of mental illness, current psychological assessment does not meet transplantation criteria.
6. Other situations where the organ transplant physician assesses the patient as not suitable for transplantation.
7. Poor compliance of the recipient or other situations deemed by the researcher as unsuitable for inclusion in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Muscle Relaxant Usage | During surgery (intraoperative intervals, and end of anesthesia)
  Total dosage of cisatracurium administered intraoperatively, including induction dose and supplemental doses.

SECONDARY OUTCOMES:
Intraoperative Sedative and Analgesic Drug Usage | During surgery (intraoperative intervals, and end of anesthesia)
  Total amount of sedatives (e.g., propofol, dexmedetomidine) and analgesics (e.g., remifentanil, sufentanil).
Anesthetic Depth (BIS Monitoring) | During surgery (intraoperative intervals, and end of anesthesia)
  Bispectral Index (BIS) values to assess adequacy of anesthetic depth, 0-40: Deep sedation or unconscious state (e.g., maintenance phase of general anesthesia); 40-60: Ideal range for general anesthesia (commonly used in surgery); 60-90: Mild to moderate sedation or gradual awakening; 90-100: Fully awake.
Intraoperative Ventilation Effect | Intraoperative key time points (e.g., post-induction, during operation, end of operation)
  Arterial PaO₂:
  Normal PaO2 values: 80-100 mmHg PaO2 60-80 mmHg: Mild hypoxia PaO2 45-60 mmHg: Moderate hypoxia PaO2 < 45 mmHg: Severe hypoxia
  Arterial PaCO₂:
  PaCO₂ 35-45 mmHg, normal value PaCO₂ < 35 mmHg, hypocapnia PaCO₂ > 45 mmHg, hypercapnia
Intraoperative Hemodynamic Stability | During surgery (intraoperative intervals, and end of anesthesia)
  Invasive arterial pressure variability/Blood pressure fluctuations at key time points
Operation and Anesthesia Duration | During surgery (intraoperative intervals, and end of anesthesia)
  This outcome measure is primarily used to record the duration of surgery and anesthesia for each patient, and to compare whether the two anesthesia methods affect the surgical process.
Postoperative Awakening and Recovery Time | Perioperative/Periprocedural
  Time to awakening and recovery of consciousness sufficient for extubation/LMA removal. From end of anesthesia to extubation/LMA removal
Perioperative Pain Scores | up to 24 hours post operatively
  Visual Analog Scale (VAS) Score range: 0-10, a score of 0 indicates no pain, while a higher score indicates a greater degree of pain.
  Prince-Henry Score (thoracoabdominal pain) Score range: 0-4 0: No pain when coughing
  1. Pain when coughing
  2. No pain at rest, pain when taking deep breaths
  3. Mild pain at rest, tolerable
  4. Severe pain at rest, unbearable
Postoperative Pulmonary Complications | From intraoperative to three months postoperatively
  Hypoxemia, Atelectasis, Pneumonia, Respiratory distress, etc.
Non-Pulmonary Complications | From intraoperative to three months postoperatively
  Hoarseness, Vocal cord paralysis, Nausea/vomiting, Arrhythmia, Delirium, etc.
Serum creatinine | Postoperative day 1-90
  Unit: μmol/L
Estimated GFR | Postoperative day 1-90
  Male Ccr = [(140 - age) × weight (kg)] / [0.818 × Scr (umol/L)] Female Ccr = [(140 - age) × weight (kg)] / [0.818 × Scr (umol/L)]*0.85
Urine output | up to 7 day post operatively
  24-hour total urine output